CLINICAL TRIAL: NCT03416114
Title: RegistRare: a Retro-prospective Registry of Rare Primary Headaches in Italian Tertiary
Brief Title: RegistRare: a Retro-prospective Registry of Rare Primary Headaches in Italian Tertiary Headache Centres
Acronym: RegistRare
Status: Recruiting | Type: Observational
Sponsor: Silvia Benemei (Other)
Collaborators: University of Modena and Reggio Emilia (Other); University of Roma La Sapienza (Other); University of Naples (Other); University of Trieste (Other); Maggiore Bellaria Hospital, Bologna (Other); University of L'Aquila (Other)
Responsible Party: Sponsor-Investigator, Silvia Benemei, Researcher, University of Florence
Organization: University of Florence (Other)
Other Study IDs: RegistRare
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Headache Disorders
Keywords: rare headaches; epidemiology
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retro-prospective survey on specific and overall prevalence and incidence of rare primary headaches (Part One, Chapter 3 and Chapter 4, ICHD-3 beta) in patients referred to Italian Tertiary Headache Centres in a 3-year (May 1, 2014-April 30, 2017 - retrospective data) and annually (from May 1, 2017 - prospective data).

DETAILED DESCRIPTION:
We planned to collect data from May 1, 2014 and afterwards, by means of both retrospective and prospective approaches.

All patients who have received or will receive a diagnosis of rare primary headache will be asked to participate and, to this aim, to give their informed consent. Each participating Centre should have received the approval of the competent Ethics Committee before commencing any study procedures.

The registry will contain anagraphic information and data about diagnosis, treatment, comorbidity, and clinical features of the headache. Patients' data will be coded through the Italian Health System unique identifier, in order to avoid duplications of patients referring to more than one Centre and also to monitor multiple referrals.

A web-based open source platform (SurveyMonkey.org) will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rare primary headaches (Part One, Chapter 3 and Chapter 4, ICHD-3 beta)
* signed informed consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data collection:
  Patients referred to Italian Tertiary Headache Centres in a 3-year (May 1, 2014 to April 30, 2017) period
  Prospective data collection:
  Patients referred to Italian Tertiary Headache Centres after April 30, 2017
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and prevalence in Tertiary headache Centres | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Benemei, MD, Study Chair — Careggi University Hospital
Locations (1):
- Careggi University Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lupi C, Evangelista L, Favoni V, Granato A, Negro A, Pellesi L, Ornello R, Russo A, Cevoli S, Guerzoni S, Benemei S. Rare primary headaches in Italian tertiary Headache Centres: Three year nationwide retrospective data from the RegistRare Network. Cephalalgia. 2018 Jul;38(8):1429-1441. doi: 10.1177/0333102418768824. Epub 2018 May 12. PMID 29754500